CLINICAL TRIAL: NCT03467516
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Adoptive Transfer of Autologous Tumor Infiltrating Lymphocytes in Patients With Metastatic Uveal Melanoma
Brief Title: Adoptive Transfer of Tumor Infiltrating Lymphocytes for Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Udai Kammula (Other)
Responsible Party: Sponsor-Investigator, Udai Kammula, Director, Solid Tumor Cell Therapy Program, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 17-219
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Uveal Neoplasms; Melanoma, Uveal
Keywords: Metastatic Uveal Melanoma; Uveal Diseases; Melanoma
MeSH Terms: conditions — Uveal Neoplasms; Uveal Melanoma; Uveal Diseases; Melanoma

STUDY DESIGN:
Intervention Model Description: The Phase 2 study will follow the Simon's optimal two-stage design. Fifteen patients will be included in the first stage; if there are 1 or fewer patients responding to therapy the trial will be terminated. If at least 2 responses are observed, expansion into Stage 2 to a total of 47 patients will occur. If at least 6 patients respond to therapy, the study therapy would be considered to have met its primary study goal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tumor Infiltrating Lymphocytes (TIL) (Experimental): Patients with uveal melanoma will receive the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide followed by infusion of up to 2x10^11 TIL infused intravenously through a central vein catheter and Aldesleukin, administered at a dose of 600,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period approximately every 8 hours beginning within 24 hours of TIL infusion and continuing for up to a maximum of 6 doses.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — TIL infusion intravenously through a central vein catheter over 20-30 minutes. Folowed by Aldesleukin, administered at a dose of 600,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period approximately every 8 hours beginning within 24 hours of TIL infusion and continuing for up to a maximum of 6 doses.

SUMMARY:
This is a Phase 2 study in which the efficacy of a non-myeloablative lymphodepleting preparative regimen followed by infusion of autologous TIL and high-dose aldesleukin in patients with metastatic uveal melanoma will be evaluated.

Metastatic uveal melanoma (UM) carries a poor prognosis with estimated survival of 4-6 months. There are no known effective systemic therapies. Metastatic UM is classified as an "orphan" disease and there are currently few clinical trial options for these patients. Thus, novel systemic approaches are desperately needed.

A recent pilot study has found that administration of autologous tumor infiltrating lymphocytes (TIL) generated from resected metastases can induce objective tumor response and durable complete response in metastatic uveal melanoma patients. These encouraging results require confirmation to determine if this immunotherapy is of future benefit in treating this disease.

DETAILED DESCRIPTION:
STUDY DESIGN

The Phase 2 study will be conducted in conjunction with companion protocol (Cell Harvest and Preparation to Support Adoptive Cell Therapy Clinical Protocols and Pre-Clinical Studies) as described below:

Cell Preparation:

Patients with evaluable metastatic uveal melanoma who have lesions that can be resected with minimum morbidity will undergo resection of tumor. TIL will be obtained while enrolled on the companion protocol (Cell Harvest and Preparation to Support Adoptive Cell Therapy Clinical Protocols and Pre-Clinical Studies). Separate tumor procurements may be performed under a protocol to obtain TIL if initial tumor procurements could not successfully generate TIL. The TIL will be grown and expanded for this trial according to standard operating procedures submitted in the IND. The TIL will be assessed for potency by interferon-gamma release.

Treatment Phase:

Once cells exceed the potency requirement and are projected to exceed the minimum number specified in the COA, the patient will be registered on this study and receive the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide, followed by infusion of up to 2x10^11 lymphocytes (minimum of 1x10^9 cells) and administration of high-dose intravenous aldesleukin. It is anticipated that TIL that meet the COA will not be achievable in approximately 20% of patients who undergo resection. These patients may undergo a second resection to grow TIL, if another suitable lesion exists. Approximately 6 weeks (+/- 2 weeks) after TIL administration, patients will undergo a complete tumor evaluation and evaluation of toxicity and immunologic parameters. Patients will receive one course of treatment. The start date of the course will be the start date of the chemotherapy; the end date will be the day of the first post-treatment evaluation. Patients may undergo a second treatment. Patients will receive no other experimental agents while on this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Measurable metastatic uveal melanoma.
* Patients must be co-enrolled on the companion protocol HCC 17-220 (Cell Harvest and Preparation to Support Adoptive Cell Therapy Clinical Protocols and Pre-Clinical Studies) and have available TIL cultures for therapy.
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* Greater than or equal to 18 years of age and less than or equal to age 75
* Able to understand and sign the Informed Consent Document
* Clinical performance status of ECOG 0 or 1
* Life expectancy of greater than three months
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the treatment.
* Serology:

  * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
* Hematology

  * Absolute neutrophil count greater than 1000/mm3 without the support of filgrastim
  * WBC ≥ 3000/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin > 8.0 g/dl
* Chemistry

  * Serum ALT/AST ≤ to 3.5 times the upper limit of normal
  * Serum creatinine ≤ to 1.6 mg/dl
  * Total bilirubin ≤ to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a clinically manageable level (except for toxicities such as alopecia or vitiligo). (Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less)

Exclusion Criteria:

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Active systemic infections (e.g.: requiring anti-infective treatment), coagulation disorders or any other active major medical illnesses.
* History of clinically significant major organ autoimmune disease
* Concurrent systemic steroid therapy.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* History of active coronary or ischemic symptoms.
* Documented LVEF of less than or equal to 45%; note: testing is required in patients with:

  * Age > 65 years old
  * Clinically significant atrial and or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or have a history of ischemic heart disease, chest pain.
* Documented FEV1 less than or equal to 60% predicted tested in patients with:

  * A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
  * Symptoms of respiratory dysfunction
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Post TIL infusion, up to 24 months (measurements taken at 6 weeks, 12 weeks, 6 months, 9 months, 12 months, 18 months 24 months)
  The proportion of patients with response per RECIST for a (minimum) time period.
  Equation: #patients with CR + #patients with PR / #patients with CR + #patients with PR + #patients with SD + #patients with PD

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | : Post TIL infusion up to 24 months (measurements taken at 6 weeks, 12 weeks, 6 months, 9 months, 12 months, 18 months 24 months)
  The proportion of patients with complete response per RECIST for a (minimum) time period.
  Equation: #patients with CR / #patients with CR + #patients with PR + #patients with SD + #patients with PD
Duration of Response (DOR) | Up to 24 months
  Time between the initial response to treatment per RECIST and subsequent disease progression (Median 'time to progression' (months) among patients achieving CR or PR).
Disease Control Rate (DCR) | Post TIL infusion up to 24 months (measurements taken at 6 weeks, 12 weeks, 6 months, 9 months, 12 months, 18 months 24 months)
  The proportion of patients with response or stable disease per RECIST for a (minimum) time period. Equation: # patients with CR + # patients with PR + # patients with SD / # patients with CR + # patients with PR + # patients with SD + # patients with PD
Progression Free Survival (PFS) | Post TIL infusion up to 24 months (measurements taken at 6 weeks, 12 weeks, 6 months, 9 months, 12 months, 18 months 24 months)
  The length of time after TIL infusion that a patient lives with the disease but it does not get worse.
Overall Survival (OS) | Post TIL infusion up to 24 months (measurements taken at 6 weeks, 12 weeks, 6 months, 9 months, 12 months, 18 months 24 months)
  The length of time from the start of treatment that patients are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Udai S Kammula, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No